CLINICAL TRIAL: NCT06739460
Title: Comparison of Antinociceptive Effects of Ketamine and Magnesium Used for Sedation in Hysteroscopy Cases
Status: Enrolling by invitation | Type: Observational
Sponsor: SULEYMAN SARI (Other Government)
Responsible Party: Sponsor-Investigator, SULEYMAN SARI, Attending Physician, Ankara Etlik City Hospital
Organization: Ankara Etlik City Hospital (Other Government)
Other Study IDs: AEŞH-EK1-2024-0056
Record Dates: First submitted 2024-11-26; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Hysteroscopy
Keywords: Magnesium; Sedation; Hysteroscopi; Opioid; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- P group: This group consists of hysteroscopy cases in which sedation was given using fentanyl, midazolam, propofol and remifentanil.
- K group: This group consists of hysteroscopy cases in which sedation was given using fentanyl, midazolam, ketamine, propofol and remifentanil.
- KM group: This group consists of hysteroscopy cases that received preoperative magnesium sulfate and sedation using fentanyl, midazolam, ketamine, propofol and remifentanil.

SUMMARY:
This study aims to compare the antinociceptive effects of ketamine and magnesium used in addition to midazolam, fentanyl, propofol and remifentanil agents preferred in hysteroscopy cases. It is conducted to observe the effect of ketamine and magnesium use on total additional propofol doses and additional remifentanil doses.

DETAILED DESCRIPTION:
Sedation is generally preferred in hysteroscopy cases. The most commonly used intravenous drugs are midazolam, fentanyl, propofol and remifentanil. Multimodal analgesia, which is intended to be provided in hysteroscopy cases, is a strategy that includes the use of two or more analgesic agents and techniques to provide adequate analgesia; and aims to minimize side effects such as bradycardia, hypotension, respiratory depression, pruritus, and postoperative nausea and vomiting. Multimodal analgesia improves patient and surgical comfort by applying additional drugs to existing agents, reduces postoperative complications, and thus helps to shorten hospital stays and reduce costs. Whether magnesium contributes to this multimodal analgesia will be investigated observationally, based on its antinociceptive effects.

ELIGIBILITY:
Inclusion Criteria:

1. ASA I-II patients
2. Patients aged 18-55
3. Patients undergoing hysteroscopy

Exclusion Criteria:

1. Patients who develop surgical complications during hysteroscopy
2. Patients with cardiovascular failure (ejection fraction <40%, patients with atrioventricular conduction disorder
3. Patients with history of cerebrovascular disease
4. Liver dysfunction (transaminases above normal level), Renal failure (creatine > 150 μmol/L),
5. Preoperative opioid use
6. History of neuromuscular disease
7. History of drug or alcohol abuse
8. Patients who develop the need for endotracheal intubation

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients receiving sedation for gynecological hysteroscopic surgery in the gynecology operating room of Ankara Etlik City Hospital
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Antinociceptive effects of ketamine and magnesium | During the hysteroscopic procedures.
  Observe the effect of ketamine and magnesium use on total additional doses of propofol and additional doses of remifentanil.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Telci L, Esen F, Akcora D, Erden T, Canbolat AT, Akpir K. Evaluation of effects of magnesium sulphate in reducing intraoperative anaesthetic requirements. Br J Anaesth. 2002 Oct;89(4):594-8. doi: 10.1093/bja/aef238. PMID 12393361
- [Background] Gao PF, Lin JY, Wang S, Zhang YF, Wang GQ, Xu Q, Guo X. Antinociceptive effects of magnesium sulfate for monitored anesthesia care during hysteroscopy: a randomized controlled study. BMC Anesthesiol. 2020 Sep 21;20(1):240. doi: 10.1186/s12871-020-01158-9. PMID 32957926
- [Background] Shin HJ, Na HS, Do SH. Magnesium and Pain. Nutrients. 2020 Jul 23;12(8):2184. doi: 10.3390/nu12082184. PMID 32718032